CLINICAL TRIAL: NCT02012010
Title: Comparison of Manual Syringe Infusion Method and Conventional Pump Infusion Method for Hysteroscopic Procedures: a Randomized Controlled Trial.
Brief Title: Comparison of Infusion Methods for Hysteroscopic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 102124-F
Record Dates: First submitted 2013-12-06; First posted 2013-12-16 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Complication of Surgical Procedure
Keywords: hysteroscopy, water intoxication, hyponatremia
MeSH Terms: conditions — Water Intoxication; Hyponatremia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual syringe infusion method (Experimental): Infuse the distension medium of hysteroscopy by manual syringe infusion method
  Interventions: Procedure: Manual syringe infusion method
- Pump infusion method (Active Comparator): Infuse the distension medium of hysteroscopy by pump infusion method
  Interventions: Procedure: Pump infusion method

INTERVENTIONS:
Procedure: Manual syringe infusion method — Infuse the distension medium of hysteroscopy by manual syringe infusion method
  Arms: Manual syringe infusion method
Procedure: Pump infusion method — Infuse the distension medium of hysteroscopy by pump infusion method
  Arms: Pump infusion method

SUMMARY:
This study is to perform a randomized controlled trial of comparing the manual syringe infusion method with the conventional pump infusion method to clarify if the manual syringe infusion method really needs less amount of distension medium.

DETAILED DESCRIPTION:
Hysteroscopy is frequently used for diagnosing abnormal uterine bleeding, endometrial polyp or submucous myoma. However, hysteroscopic procedure can cause morbidity and even mortality related to infusion distension medium. We had used a manual syringe infusion method to infuse fluid for distending the uterine cavity in our institute without significant morbidity, and it seems that this method need less amount of distension medium, and possible result in less possibility of hyponatremia. Therefore, the aim of this study is to perform a randomized controlled trial of comparing the manual syringe infusion method with the conventional infusion pump method to clarify if the manual syringe infusion method really needs less amount of distension medium during hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Of greater than twenty-year-old female patients suffering from abnormal uterine bleeding, suspected endometrial lesions, endometrial polyp, or submucous myoma.

Exclusion Criteria:

* Female patients of less than twenty years-old.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-12-06 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
The difference in the amount of distension medium used | 1 day
  The amount of distension medium used between the manual syringe infusion method and the conventional infusion pump method of hysteroscopic surgery

SECONDARY OUTCOMES:
The difference of serum sodium and pain score, operation time | 1 day
  The difference of serum sodium and pain score, operation time between these two distension medium infusion methods of hysteroscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Mou Hsiao, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan